CLINICAL TRIAL: NCT07193108
Title: The 30-15 Intermittent Fitness Test Provides Superior Sport-Specific Sensitivity to Treadmill Testing in Elite Female Footballers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gümüşhane Universıty (Other)
Responsible Party: Principal Investigator, Coşkun YILMAZ, ASSOC. PROF., Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025-0451
Record Dates: First submitted 2025-09-12; First posted 2025-09-25 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Change in Maximal Oxygen Uptake (VO₂Max)
Keywords: aerobic capacity; intermittent fitness assessment; women's football; metabolic response

STUDY DESIGN:
Intervention Model Description: This study used a randomized crossover design in which all participants completed both the 30-15 Intermittent Fitness Test and a treadmill-based incremental running test. The order of the test protocols was randomized, and a 48-hour recovery period was implemented between sessions to minimize carryover effects. Physiological responses were compared within participants across the two testing conditions.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30-15 Intermittent Fitness Test (30-15IFT) (Experimental): Participants performed the 30-15 Intermittent Fitness Test consisting of 30-second running bouts interspersed with 15-second passive recovery periods, with progressive increases in running speed until volitional exhaustion.
  Interventions: Other: 30-15 Intermittent Fitness Test; Other: Control
- CONTROL (No Intervention): Inspiratory Muscle Warm-Up Non-treated group, Control

INTERVENTIONS:
Other: 30-15 Intermittent Fitness Test — Participants performed the 30-15 Intermittent Fitness Test consisting of 30-second running bouts interspersed with 15-second passive recovery periods, with progressive increases in running speed until volitional exhaustion.
  Arms: 30-15 Intermittent Fitness Test (30-15IFT)
Other: Control — Inspiratory Muscle Warm-Up Non-treated group, Control
  Arms: 30-15 Intermittent Fitness Test (30-15IFT)

SUMMARY:
This study compares the acute aerobic, metabolic, and threshold-related physiological responses elicited by the 30-15 Intermittent Fitness Test (30-15IFT) and a treadmill-based incremental running test in elite female football players. Using a randomized crossover design, all participants completed both testing protocols with a 48-hour recovery period. Outcomes included maximal oxygen uptake, maximal running speed, heart rate responses, lactate-derived thresholds, metabolic tolerance indices, and recovery markers.

DETAILED DESCRIPTION:
Laboratory-based treadmill tests are commonly used to assess aerobic capacity in football players; however, they lack sport-specific characteristics such as intermittent running, accelerations, and changes of direction. The 30-15 Intermittent Fitness Test (30-15IFT) has been proposed as a more ecologically valid field-based alternative.

Twenty-seven elite female football players competing in the Turkish Women's Super League completed both the 30-15IFT and a standardized treadmill incremental protocol in a randomized crossover design. Tests were separated by 48 hours and performed under controlled environmental conditions. Physiological variables including VO₂max, maximal running speed, maximal heart rate, respiratory exchange ratio, lactate-derived thresholds (OBLA), metabolic load-dependent tolerance, and post-exercise recovery markers were assessed using breath-by-breath gas analysis, heart rate monitoring, and capillary blood lactate sampling.

The study aims to determine whether the 30-15IFT elicits more sensitive and sport-specific physiological responses compared with treadmill testing, thereby supporting its use in performance monitoring and individualized training prescription in elite women's football.

ELIGIBILITY:
Inclusion Criteria:

* Female football players aged 18-35 years
* Competing in the Turkish Women's Super League
* Minimum of 3 years of professional football experience,
* Full participation in training and matches during the previous 6 months,
* Ability to perform maximal exercise testing

Exclusion Criteria:

* Musculoskeletal injury affecting performance within the last 3 months,
* Diagnosed cardiovascular, metabolic, or respiratory disease,
* Any condition limiting maximal physical effort

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Maximal Running Speed (MRS) | DAY 1
  Highest running speed achieved during each protocol.
Maximal Oxygen Uptake (VO₂max) | Day 1
  Maximal oxygen uptake measured via breath-by-breath gas analysis.

SECONDARY OUTCOMES:
body composition | 1 Day
  Body composition (BMI)
Maximal Heart Rate (HRmax) | 1 Day
  Peak heart rate achieved during each test.
Maximal Oxygen Uptake (VO₂max) | DAY 1
  Maximal oxygen uptake measured via breath-by-breath gas analysis.

CONTACTS AND LOCATIONS:
Overall Officials: coşkun yılmaz, associate professor, Principal Investigator — Gümüşhane Universıty
Locations (1):
- Gumushane Univetsity, Gümüşhane, Kelkit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol